CLINICAL TRIAL: NCT04173988
Title: A Single Center, Open Label, Single Arm Exploratory Clinical Study of CD19-Directed Allogeneic Chimeric Antigen Receptor CART-cell Immunotherapy Cell Therapy in Pediatric Patients With Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Study of alloCART-19 Cell Therapy in Pediatric Patients With Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xiaowen Zhai, vice president, Children's Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-272
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: ALL, Childhood B-Cell
Keywords: Allogeneic CAR-T19
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- alloCART-19 (Experimental): For the very first patient, the initial dose could be administered via one or three intravenous infusions within 1 to 5 days. Starting from the second patient, the investigator will decide whether to use single or multiple alloCART-19 infusions, based on the treatment experience at previous dose level(s) and the patient's baseline disease burdens.
  A lymphodepletion conditioning with cyclophosphamide and fludarabine will be conducted before alloCART-19 infusion.
  Interventions: Genetic: alloCART-19; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Genetic: alloCART-19 — AlloCART-19 is an allogeneic CAR-T cell product targeting CD19.
  * For children with body weight ≤ 50 kg, dose range for dose escalation will be 0.5 - 5 × 10^6 CAR+ cells/kg
  * For children with body weight > 50 kg, dose range for dose escalation will be 0.25 - 2.5 × 10^8 CAR+ cells.
  Other Names: allogeneic CAR-T19
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion
  Other Names: no other intervention names
Drug: Fludarabine — Chemotherapy for lymphodepletion
  Other Names: no other intervention names

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of CD19-Directed Allogeneic Chimeric Antigen Receptor T- cell (alloCART-19)therapy in pediatric patients with relapsed/refractory acute lymphoblastic leukemia（ALL）.

DETAILED DESCRIPTION:
This is a single center, open label, single arm, dose escalation study to explore the safety, tolerability, and pharmacokinetic / pharmacodynamic profile of CD19-Directed Allogeneic Chimeric Antigen Receptor T- cell (alloCART-19) in pediatric patients with relapsed or refractory B-cell acute lymphoblastic leukemia. The study will also assess the preliminary efficacy of CD19-Directed Allogeneic Chimeric Antigen Receptor T- cell (alloCART-19). For this exploratory clinical trial, approximately 3-6 patients will be enrolled. During dose escalation, at least one evaluable patient will be enrolled at each dose level. Once DLT is reached, 1 to 3 additional patients will be enrolled at the dose level below DLT, which has been tested and determined to be safe in the trial, to evaluate the optimal safe and therapeutic dose to be approved by the investigator and sponsor.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent and assent forms if applicable must be obtained prior to the start of any research procedure
* Age 1 year at the time of screening to age 18 years at the time of initial diagnosis
* Relapsed/refractory pediatric ALL that meet one of the following conditions:

  1. Incomplete patients with conventional chemotherapy regimens, or primary refractory patients who failed to complete remission with 2 courses of standard chemotherapy regimen, or did not achieve complete remission after first-line or multi-line salvage chemotherapy
  2. Early recurrence after complete remission (< 12 months) or late recurrence after complete remission (≥ 12 months) and chemotherapy was not completely relieved by the standardized two course induction regimens
  3. Recurrence after autologous or allogeneic hematopoietic stem cell transplantation
* Patients who are Philadelphia chromosome-positive (Ph+) are eligible if they have failed at least 2 lines of chemotherapy and have failed two lines of TKI therapy or if TKI therapy is contraindicated.
* For relapsed patients, CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry within 3 months of study entry
* Karnofsky performance status of > 60 at screening
* During the screening period and within 10 days of treatment, adequate organ function defined as:

  1. Renal Function: serum creatinine ≤ 2 x ULN
  2. Liver Function: ALT and/or AST ≤ 10 x ULN (depending on age), bilirubin ≤ 5 x ULN
  3. Pulmonary Function: oxygen saturation ≥ 91%
  4. Heart Function: echocardiogram (ECHO): left ventricular ejection fraction (LVEF) ≥ 45%
* Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening or immunological/molecular biological results with persistent MRD
* Female subjects of childbearing age must have a negative serum or urine pregnancy test during the screening period and agree to take effective contraceptive measures during the trial period until the last follow-up

Exclusion Criteria

* Pregnant or lactating women
* Unable to tolerate venipuncture
* Prior history of:

  1. Allogeneic cell therapy (including hematopoietic stem cell transplantation) within 6 weeks of alloCART-19 infusion
  2. Any live vaccine within 4 weeks of alloCART-19 infusion and/or plan to receive live vaccine after enrollment
  3. Immunosuppressants for GvHD treatment within 4 weeks of alloCART-19 infusion
  4. Systemic corticosteroid treatment at doses greater than 5 mg/day prednisone*3 days (or equivalent corticosteroids) within 72 hours prior to alloCART-19 treatment
  5. Before receiving alloCART-19 treatment, had received the following anti-neoplastic therapies: Tyrosine kinase inhibitors and hydroxyurea within 72 hours; Vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate < 25 mg/m2, cytosine arabinoside < 100 mg/m2/day, or asparaginase (non-pegylated) within 1-week; Pegylated-asparaginase within 4 weeks; Central nervous system disease prophylaxis (e.g. intrathecal methotrexate) within 1 week; Investigational drug treatment within 4 weeks
  6. Had received the following anti-neoplastic radiotherapy before receiving alloCART-19 treatment: Radiotherapy for non-CNS sites within 2 weeks; Radiotherapy for the CNS site within 8 weeks
* Have the following medical history:

  1. Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD)
  2. Isolated extramedullary disease recurrence (e.g. central nervous system and testis)
  3. Previous or active central nervous system (CNS) diseases such as seizures, cerebral ischemia/bleeding, dementia, cerebellar disease or any autoimmune disease involving CNS
  4. Previous malignant tumors (excluding curative trends and inactive skin cancer in situ or cervical cancer)
  5. Genetic syndromes associated with bone marrow failure states: such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome (excluding Down syndrome)
  6. Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening period)
  7. History of HIV, or HIV-positive test within 8 weeks of screening period
  8. Any uncontrolled serious infection during the screening period
  9. Severe, poorly controlled concomitant diseases such as, but not limited to, nervous system, kidney, liver, endocrine or gastrointestinal disorders that may be deemed by the investigator to interfere with the inclusion of the subject in the study.
  10. Any clinical abnormalities including but not limited to the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism and bones that may be deemed by the investigator to interfere with the inclusion of a subject in the study.
* The following treatments and/or medications must be excluded:

  1. Simultaneous application of other anti-neoplastic drugs, including traditional Chinese herbal medicines
  2. Drugs that prolong the QT interval (including Ia and III antiarrhythmic drugs)
  3. Daily oxygen therapy
  4. long-term use of corticosteroids (except for inhaled and topical use)
* Any circumstance or condition that in the judgement of the investigator may interfere with the subject's participation in the trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Day 28 after the first alloCART-19 infusion
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality per Lee DW and Locke FL standards and management guideline, and should be possibly related to alloCART-19 cell therapy, and should be unrelated to the disease itself, disease progression, concomitant diseases or concomitant medication. DLT will be analyzed as categorical variable，coded as 1 for DLT occur, 0 for no DLT.

SECONDARY OUTCOMES:
The occurrence of adverse events | After the first alloCART-19 infusion for 2 year
  The adverse events (AE) is a composite variable including liver and kidney function damage, nausea, vomiting, arrhythmia and dyspnea. The variable would be coded as 1 if any of these events occurs after the first alloCART-19 infusion while 0 for none . These adverse events would be measured by assessment scale method according to NCI CTC AE v5.0 classification standard.
Objective Response Rate | Day 28 and 3 months after the first alloCART-19 infusion
  Objective Response Rate（ORR）is defined as the proportion of patients whose tumor volume shrank to a predetermined value and the minimum time limit required.
  ORR = complete remission (CR) + incomplete complete remission (CRi)
Best Overall Response | Day 28 and 3 months after the first alloCART-19 infusion
  Best Overall Response（BOR）at 28 days and 3 months after drug infusion was evaluated to preliminarily evaluate the optimal efficacy of alloCART-19 infusion in patients.

OTHER OUTCOMES:
AlloCART-19 cells | After the first alloCART-19 infusion for 2 years
  AlloCART-19 cells would be detected in peripheral blood, bone marrow, and/or CSF.
  The variable would be coded as 1 if any alloCART-19 cell was founded in the tissues metioned above while 0 for none.
T cell subsets | After the first alloCART-19 infusion for 2 years
  T cell subsets is a composite varible including CD3, CD4 and CD8 ratio observed in blood and bone marrow. The variable would be coded as 1 if any of these observations were not in normal range while 0 for all normal.

CONTACTS AND LOCATIONS:
Overall Officials: zhai xiaowen, PhD, Study Director — PI
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Minhang, China

IPD SHARING:
Plan to Share IPD: No